CLINICAL TRIAL: NCT02591420
Title: Safety and Virologic Effect of a Human Monoclonal Antibody, VRC-HIVMAB060-00-AB (VRC01), With Broad HIV-1 Neutralizing Activity, Administered Intravenously to Adults During Early Acute HIV Infection
Brief Title: Safety and Virologic Effect of a Human Monoclonal Antibody (VRC01) Administered Intravenously to Adults During Early Acute HIV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RV 398; 12002 (Registry Identifier: DAIDS-ES); WRAIR 2166 (Other: NIAID)
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — VRC01 monoclonal antibody

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: immediate ART and placebo infusion (Experimental): Participants will start ART and will receive a single infusion of placebo at Day 0.
  Interventions: Biological: Placebo for VRC01; Drug: Antiretroviral therapy (ART) (regimen will vary within countries and by patient)
- Group 2: immediate ART and VRC01 infusion (Experimental): Participants will start ART and receive a single infusion of VRC01 at Day 0.
  Interventions: Biological: VRC01; Drug: Antiretroviral therapy (ART) (regimen will vary within countries and by patient)
- Group 3: immediate VRC01 infusion and subsequent ART (Experimental): Participants will receive a single infusion of VRC01 on Day 0 followed by ART initiation on Day 7.
  Interventions: Biological: VRC01; Drug: Antiretroviral therapy (ART) (regimen will vary within countries and by patient)

INTERVENTIONS:
Biological: VRC01 — 40 mg/kg of VRC01 will be administered as an intravenous infusion over 30 to 60 minutes using a volumetric pump
  Other Names: VRC-HIVMAB060-00-AB
  Arms: Group 2: immediate ART and VRC01 infusion; Group 3: immediate VRC01 infusion and subsequent ART
Biological: Placebo for VRC01 — Administered as an intravenous infusion over 30 to 60 minutes using a volumetric pump
  Arms: Group 1: immediate ART and placebo infusion
Drug: Antiretroviral therapy (ART) (regimen will vary within countries and by patient) — ART is provided by the study sites and consists of country guideline-recommended, available first line once-daily oral combination therapy: currently either efavirenz 600 mg/emtricitabine 200 mg/tenofovir disoproxil fumarate 300 mg or efavirenz 600 mg/lamivudine 300 mg/tenofovir disoproxil fumarate 300 mg. This initial ART regimen may be adjusted or switched to an alternate regimen as clinically indicated for regimen intolerance or failure.

SUMMARY:
This study will evaluate the safety and virologic effect of an experimental human monoclonal antibody (mAb), VRC-HIVMAB060-00-AB (VRC01), alone or in combination with antiretroviral therapy (ART), in adults during early acute HIV infection.

DETAILED DESCRIPTION:
Human monoclonal antibodies (mAbs) may have the potential to treat HIV infection by preventing the spread of the virus. This study will evaluate an experimental mAB known as VRC-HIVMAB060-00-AB (VRC01). The purpose of this study is to evaluate the safety and virologic effect of VRC01, alone or in combination with ART, in adults with early acute HIV infection. Researchers will also evaluate the effect of VRC01 on the establishment of an HIV reservoir during early acute HIV infection.

This study will enroll participants who are diagnosed with early acute HIV infection. Participants will be randomly assigned to one of three groups: Group 1 will begin ART and receive a single infusion of placebo at Day 0. Group 2 will begin ART and receive a single infusion of VRC01 at Day 0. Group 3 will receive a single infusion of VRC01 on Day 0 and begin ART on Day 7. ART will vary by country and will consist of country guideline-recommended, available first line combination therapy: currently either efavirenz 600 mg/emtricitabine 200 mg/tenofovir disoproxil fumarate 300 mg or efavirenz 600 mg/lamivudine 300 mg/tenofovir disoproxil fumarate 300 mg. This initial ART regimen may be adjusted or switched to an alternate regimen as clinically indicated for regimen intolerance or failure.

Study visits will occur at Days 0, 1, 3, 7, 10, 14, 18, 21, 25, 28, 42, 56, 84, 112, 168, and 175. Visits will include a physical examination, medical history review, and blood collection. Neurocognitive testing will take place on Day 168. Some participants may take part in optional study procedures at various time points during the study including mucosal secretion collection, rectosigmoid biopsy, lymph node biopsy, leukapheresis, and lumbar puncture.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to complete the informed consent process
* Passes Test of Understanding
* 18 to 50 years of age
* Experiencing early acute HIV-1 infection as defined by blood samples on at least two separate days positive by nucleic acid testing within 21 days of a negative nucleic acid HIV-1 test OR by a positive nucleic acid test or a positive 4th generation enzyme immunoassay (EIA) in the context of a negative 2nd or negative 3rd generation HIV EIA test
* No history of antiretroviral therapy for any indication in the last 30 days.
* In general good health
* Willing to have blood samples collected and stored
* Able to participate for 25 weeks for study visits
* Willing to have photo or fingerprint taken for identification purposes

Female-Specific Criteria:

* Agrees not to become pregnant from the time of study enrollment until the last study visit. If a woman has no history of hysterectomy, tubal ligation or menopause, she must agree to use an effective birth control method: abstinence; male or female condoms; diaphragm or cervical cap with spermicide; intrauterine device; contraceptive hormones delivered by pills, patch, injections, or vaginally; and hormonal implants under the skin; or a male partner who has previously undergone a vasectomy.
* Negative beta-human chorionic gonadotropin (HCG) pregnancy test (urine or serum) on day of enrollment for any woman unless she is post-menopause for 24 consecutive months or has undergone a surgical procedure that precludes pregnancy

Exclusion Criteria:

* Weight less than 46 kg or greater than 115 kg
* Previous receipt of humanized or human monoclonal antibody whether licensed or investigational
* Ongoing AIDS-related opportunistic infection (including oral thrush or active tuberculosis)
* Severe acute retroviral syndrome (as defined in Appendix I of the protocol) or clinical condition (other than HIV infection) constituting an indication for immediate antiretroviral therapy per local country guidelines
* Active injection drug use within previous 12 months
* History of a severe allergic reaction with generalized urticaria, angioedema, or anaphylaxis in the 2 years prior to enrollment
* History of chronic urticaria
* Physical finding on examination considered indicative of significant disease such as murmur (other than functional), hepatosplenomegaly, focal neurological deficit
* Hypertension that is not well controlled by medication
* Positive hepatitis B surface antigen at any time in the past
* History of hepatitis C infection
* Untreated syphilis infection
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 2 times the upper limit of normal (ULN).
* Absolute neutrophil count (ANC) less than 740 cells/mm^3
* Estimated glomerular filtration rate (GFR) less than 50 ml/min within the past 90 days
* Breastfeeding
* Pregnancy
* Receipt of licensed vaccine or other investigational study agent within 28 days prior to enrollment or past participation in an investigational HIV vaccine study with receipt of active product
* Current or planned participation in another interventional clinical trial during the study period
* Chronic or recurrent use of medications that modify host immune response, e.g., oral or parenteral steroids, cancer chemotherapy
* Any other chronic or clinically significant medical condition that in the opinion of investigator would jeopardize the safety or rights of the volunteer. Including, but not limited to: diabetes mellitus type I, chronic hepatitis, renal failure; OR clinically significant forms of: drug or alcohol abuse, mental illness, severe asthma, autoimmune disease, psychiatric disorders, heart disease, or cancer.
* Study site employee

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-04; Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LTC Julie Ake, MD, Study Chair — U.S. Military HIV Research Program (MHRP)/Henry M. Jackson Foundation for the Advancement of Military Medicine (HJF); Merlin Robb, MD, Study Chair — US Military HIV Research Program
Locations (5):
- Kenya Med. Research Inst./Walter Reed Project, Clinical Research Centre, Off Hospital Road. Kericho, Kericho, Kenya
- National Institute for Medical Research (NIMR)-Mbeya Medical Research Center (MMRC) Non-Network CRS, Mbeya, Tanzania
- Thailand (2):
  - SEARCH Thai Red Cross AIDS Research Centre Non-Network CRS, Bangkok
  - ECHO Center Non-Network CRS, Chon Buri
- Makerere University Walter Reed Project (MUWRP), Kampala, Uganda

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: Immediate ART and Placebo Infusion | Group 2: Immediate ART and VRC01 Infusion | Group 3: Immediate VRC01 Infusion and Subsequent ART
Started | 8 | 8 | 8
Completed | 8 | 7 | 6
Not Completed | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Immediate ART and Placebo Infusion | Group 2: Immediate ART and VRC01 Infusion | Group 3: Immediate VRC01 Infusion and Subsequent ART | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.9 (4.6) | 23.5 (3.2) | 24.9 (2.5) | 23.4 (3.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 6 | 4 | 4 | 14
  Gender: Female | 2 | 3 | 2 | 7
  Gender: Transgender | 0 | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 8 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 5 | 5 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 3 | 9
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Tanzania | 0 | 1 | 0 | 1
  Uganda | 1 | 0 | 1 | 2
  Kenya | 2 | 2 | 2 | 6
  Thailand | 5 | 5 | 5 | 15
Baseline Viral Load [Mean (Standard Deviation); unit: log10(copies/mL)] | 5.8115 (1.2286) | 5.6740 (0.8927) | 5.5753 (0.7120) | 5.6869 (0.9306)
Baseline CD4+ Count [Mean (Standard Deviation); unit: cells/microLiter] | 595.724 (252.350) | 500.839 (99.899) | 410.991 (158.902) | 502.518 (188.803)
Fiebig Stage [Count of Participants; unit: Participants] — Fiebig stages are: I) HIV RNA detectable, p24 antigen non-reactive, 3rd gen ELISA non-reactive; II) HIV RNA and p24 antigen detectable; 3rd gen ELISA non-reactive; III) HIV RNA and p24 antigen detectable; 3rd gen ELISA reactive, Western Blot negative; IV) HIV RNA and p24 antigen detectable; 3rd gen ELISA positive, Western Blot indeterminate; V) HIV RNA detectable, p24 antigen detectable or not detectable, 3rd gen ELISA reactive, Western Blot positive but lacking p31 band; VI) HIV RNA detectable, p24 antigen detectable or not detectable, 3rd gen ELISA reactive, Western Blot positive w/p31 band
  Participants
    Fiebig Stage 1 | 1 | 1 | 1 | 3
    Fiebig Stage 2 | 3 | 3 | 3 | 9
    Fiebig Stage 3 | 2 | 3 | 1 | 6
    Fiebig Stage 4 | 1 | 0 | 3 | 4
    Fiebig Stage 5 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 or Greater mAb-related Reactogenicity and mAb-related Adverse Events (AEs)
Description: This outcome is the combined total number of grade 3 or higher mAb-related reactogenicity events and mAb-related adverse events for each group. Only grade 3 reactogenicity events/AEs that are determined by the study physicians to be related to mAb are included. Adverse events, including reactogenicity events, are graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events v2.0 dated November 2014. This outcome is the total number of solicited adverse events (reactogenicity events) that had a severity of grade 3 or higher and were related to the mAb. Note that higher grades indicate worse severity.
Time Frame: Measured through Week 24
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Immediate ART and Placebo Infusion | Group 2: Immediate ART and VRC01 Infusion | Group 3: Immediate VRC01 Infusion and Subsequent ART
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 1

2. Primary Outcome: Plasma Viral Load Change From Day 0 to Day 7
Time Frame: Measured through Day 7
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: log(copies/mL)
Arm/Group | Group 1: Immediate ART and Placebo Infusion | Group 2: Immediate ART and VRC01 Infusion | Group 3: Immediate VRC01 Infusion and Subsequent ART
Number analyzed (Participants) | 8 | 8 | 8
log(copies/mL) | -1.5238 (0.8018) | -1.6108 (0.8174) | -0.2336 (0.9635)
Statistical Analysis 1: Comparison: Group 1: Immediate ART and Placebo Infusion vs Group 2: Immediate ART and VRC01 Infusion; Pairwise Wilcoxon rank-sum test using 10,000 bootstrapped samples; Test type: Superiority; p = .645, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 1: Immediate ART and Placebo Infusion vs Group 3: Immediate VRC01 Infusion and Subsequent ART; Test type: Superiority; p = .007, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Group 2: Immediate ART and VRC01 Infusion vs Group 3: Immediate VRC01 Infusion and Subsequent ART; Test type: Superiority; p = .003, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Time to Virologic Suppression (Less Than 50 Copies/ml) in Plasma
Time Frame: Measured through Week 24
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Group 1: Immediate ART and Placebo Infusion | Group 2: Immediate ART and VRC01 Infusion | Group 3: Immediate VRC01 Infusion and Subsequent ART
Number analyzed (Participants) | 8 | 8 | 8
Days | 58.0 [13.0 to 162.0] | 43.5 [14.0 to NA] — The upper limit of the confidence interval was not estimable because all participants considered failures for this endpoint withdrew from the study prior to reaching the <50 copies/mL threshold | 87.0 [29.0 to NA] — The upper limit of the confidence interval was not estimable because all participants considered failures for this endpoint withdrew from the study prior to reaching the <50 copies/mL threshold
Statistical Analysis 1: Comparison: Group 1: Immediate ART and Placebo Infusion vs Group 2: Immediate ART and VRC01 Infusion vs Group 3: Immediate VRC01 Infusion and Subsequent ART; Test type: Superiority; p = .347, Log Rank

4. Secondary Outcome: Number of Total Viremic Copy Days (Area Under Viral Load Curve) From Day 0 to Week 24
Time Frame: Measured through Week 24
Population: All randomized participants
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Group 1: Immediate ART and Placebo Infusion | Group 2: Immediate ART and VRC01 Infusion | Group 3: Immediate VRC01 Infusion and Subsequent ART
Number analyzed (Participants) | 8 | 8 | 8
days | 1.81 [1.44 to 2.22] | 1.74 [1.31 to 2.25] | 2.34 [1.69 to 3.18]
Statistical Analysis 1: Comparison: Group 1: Immediate ART and Placebo Infusion vs Group 2: Immediate ART and VRC01 Infusion vs Group 3: Immediate VRC01 Infusion and Subsequent ART; Test type: Superiority; p = .369, Kruskal-Wallis

5. Secondary Outcome: Measurement of Plasma Viremia Including Single Copy HIV RNA Quantification
Description: In samples with HIV RNA less than 50 copies/ml at Day 7, Day 14, and Week 24
Time Frame: Measured through Week 24
Measure: Mean (95% Confidence Interval); unit: log-10(copies/mL)
Arm/Group | Group 1: Immediate ART and Placebo Infusion | Group 2: Immediate ART and VRC01 Infusion | Group 3: Immediate VRC01 Infusion and Subsequent ART
Number analyzed (Participants) | 8 | 8 | 8
log-10(copies/mL)
  Day 7 | 4.2877 [3.7054 to 4.8906] | 4.0632 [3.5284 to 4.5666] | 5.3417 [4.9594 to 5.7843]
  Day 14 | 3.2345 [2.4737 to 3.9592] | 3.0389 [2.3121 to 3.7925] | 3.6189 [3.1457 to 4.0278]
  Week 24 (Day 168) | 0.9223 [0.7586 to 1.1457] | 0.9035 [0.7671 to 1.1079] | 0.7993 [0.6990 to 1.0000]
Statistical Analysis 1: Comparison: Group 1: Immediate ART and Placebo Infusion vs Group 2: Immediate ART and VRC01 Infusion; Comparison of groups 1 and 2 for data from day 7; Test type: Superiority; p = .645, Wilcoxon (Mann-Whitney) — p-value calculated using 10,000 bootstrap samples for day 7 data
Statistical Analysis 2: Comparison: Group 1: Immediate ART and Placebo Infusion vs Group 3: Immediate VRC01 Infusion and Subsequent ART; Comparison between groups 1 and 3 for data from day 7; Test type: Superiority; p = 0.028, Wilcoxon (Mann-Whitney) — p-value calculated using 10,000 bootstrap samples for day 7 data
Statistical Analysis 3: Comparison: Group 1: Immediate ART and Placebo Infusion vs Group 2: Immediate ART and VRC01 Infusion; Comparison of groups 1 and 2 for data from day 14; Test type: Superiority; p = 0.798, Wilcoxon (Mann-Whitney) — p-value calculated using 10,000 bootstrap samples for day 14 data
Statistical Analysis 4: Comparison: Group 1: Immediate ART and Placebo Infusion vs Group 3: Immediate VRC01 Infusion and Subsequent ART; Comparison of groups 1 and 3 for data from day 14; Test type: Superiority; p = .505, Wilcoxon (Mann-Whitney) — p-value calculated using 10,000 bootstrap samples for day 14 data
Statistical Analysis 5: Comparison: Group 1: Immediate ART and Placebo Infusion vs Group 2: Immediate ART and VRC01 Infusion; Comparison of groups 1 and 2 at study day 168 (week 24); Test type: Superiority; p > .999, Wilcoxon (Mann-Whitney) — p-value calculated using 10,000 bootstrap samples for day 168 data
Statistical Analysis 6: Comparison: Group 1: Immediate ART and Placebo Infusion vs Group 3: Immediate VRC01 Infusion and Subsequent ART; Comparison of groups 1 and 3 at study day 168; Test type: Superiority; p = 0.497, Wilcoxon (Mann-Whitney) — p-value calculated using 10,000 bootstrap samples for day 168 data

6. Secondary Outcome: Measurement of Cell-associated HIV RNA and DNA in the Peripheral Compartment
Time Frame: Measured through Week 24 (Day 168)
Population: Virologic population consists of all randomized participants.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Group 1: Immediate ART and Placebo Infusion | Group 2: Immediate ART and VRC01 Infusion | Group 3: Immediate VRC01 Infusion and Subsequent ART
Number analyzed (Participants) | 8 | 7 | 7
log10 copies/mL
  Day 0 | 4.036 (0.950) | 3.214 (1.571) | 3.940 (1.298)
  Day 3: number analyzed (Participants) | 6 | 6 | 7
  Day 3 | 3.427 (1.268) | 3.553 (0.561) | 4.090 (0.432)
  Day 7: number analyzed (Participants) | 8 | 6 | 7
  Day 7 | 3.690 (0.708) | 2.780 (0.979) | 3.924 (0.482)
  Day 28: number analyzed (Participants) | 7 | 6 | 7
  Day 28 | 2.821 (1.357) | 2.095 (1.296) | 2.823 (1.309)
  Day 168: number analyzed (Participants) | 8 | 7 | 5
  Day 168 | 2.169 (1.516) | 1.283 (1.616) | 2.656 (0.768)

7. Secondary Outcome: Percentage of Participants Experiencing Acute Retroviral Syndrome
Time Frame: Measured through Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Immediate ART and Placebo Infusion | Group 2: Immediate ART and VRC01 Infusion | Group 3: Immediate VRC01 Infusion and Subsequent ART
Number analyzed (Participants) | 8 | 8 | 8
Participants | 1 | 0 | 0

8. Secondary Outcome: Percentage of Participants Experiencing a Hospitalization
Time Frame: Measured through Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Immediate ART and Placebo Infusion | Group 2: Immediate ART and VRC01 Infusion | Group 3: Immediate VRC01 Infusion and Subsequent ART
Number analyzed (Participants) | 8 | 8 | 8
Participants | 2 | 0 | 1

9. Secondary Outcome: Percentage of Participants Experiencing Opportunistic Infections
Time Frame: Measured through Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Immediate ART and Placebo Infusion | Group 2: Immediate ART and VRC01 Infusion | Group 3: Immediate VRC01 Infusion and Subsequent ART
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

10. Secondary Outcome: Percentage of Participants Experiencing Non-AIDS-related Conditions
Time Frame: Measured through Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Immediate ART and Placebo Infusion | Group 2: Immediate ART and VRC01 Infusion | Group 3: Immediate VRC01 Infusion and Subsequent ART
Number analyzed (Participants) | 8 | 8 | 8
Participants | 8 | 7 | 7
Statistical Analysis 1: Comparison: Group 1: Immediate ART and Placebo Infusion vs Group 2: Immediate ART and VRC01 Infusion vs Group 3: Immediate VRC01 Infusion and Subsequent ART; Test type: Superiority; p > .999, Fisher Exact
Statistical Analysis 2: Comparison: Group 1: Immediate ART and Placebo Infusion vs Group 2: Immediate ART and VRC01 Infusion vs Group 3: Immediate VRC01 Infusion and Subsequent ART; This test compares group 1 to groups 2 and 3 combined (1 vs. 2 & 3); Test type: Superiority; p = 0.390, Barnard's test

11. Secondary Outcome: Measurement of CD4 + T Cells
Description: Decrease from baseline to nadir, increase from nadir to Week 24, and overall change from baseline to Week 24
Time Frame: Measured through Week 24
Population: Change is analyzed using participants with data at both time points.
Measure: Mean (95% Confidence Interval); unit: cells/microLiter
Arm/Group | Group 1: Immediate ART and Placebo Infusion | Group 2: Immediate ART and VRC01 Infusion | Group 3: Immediate VRC01 Infusion and Subsequent ART
Number analyzed (Participants) | 8 | 8 | 8
cells/microLiter
  Change from Baseline to Nadir | -84.034 [-176.61 to -14.217] | -47.206 [-99.143 to -6.206] | -42.209 [-90.054 to -5.571]
  Change from Nadir to Day 168 | 381.398 [216.101 to 561.613] | 343.764 [126.938 to 600.480] | 226.995 [97.837 to 356.153]
  Change from Baseline to Day 168 | 336.134 [118.637 to 566.003] | 333.485 [74.122 to 622.000] | 254.594 [70.404 to 380.180]
Statistical Analysis 1: Comparison: Group 1: Immediate ART and Placebo Infusion vs Group 2: Immediate ART and VRC01 Infusion; Comparison of change in CD4+ T cells in Groups 1 and 2 from baseline to Nadir; Test type: Superiority; p = 0.694, Wilcoxon (Mann-Whitney) — Comparison of change in CD4+ T cells in Groups 1 and 2 from baseline to Nadir p-value calculated using 10,000 bootstrapped samples
Statistical Analysis 2: Comparison: Group 1: Immediate ART and Placebo Infusion vs Group 3: Immediate VRC01 Infusion and Subsequent ART; Comparison of change in CD4+ T cells in Groups 1 and 3 from baseline to Nadir; Test type: Superiority; p = 0.729, Wilcoxon (Mann-Whitney); Comparison of change in CD4+ T cells in Groups 1 and 3 from baseline to Nadir p-value calculated using 10,000 bootstrapped samples
Statistical Analysis 3: Comparison: Group 1: Immediate ART and Placebo Infusion vs Group 2: Immediate ART and VRC01 Infusion; Comparison of change in CD4+ T cells in Groups 1 and 2 from Nadir to Day 168; Test type: Superiority; p = 0.694, Wilcoxon (Mann-Whitney); Comparison of change in CD4+ T cells in Groups 1 and 2 from Nadir to Day 168 p-value calculated using 10,000 bootstrapped samples
Statistical Analysis 4: Comparison: Group 1: Immediate ART and Placebo Infusion vs Group 3: Immediate VRC01 Infusion and Subsequent ART; Comparison of change in CD4+ T cells in Groups 1 and 3 from Nadir to Day 168; Test type: Superiority; p = 0.393, Wilcoxon (Mann-Whitney); Comparison of change in CD4+ T cells in Groups 1 and 3 from Nadir to Day 168 p-value calculated using 10,000 bootstrapped samples
Statistical Analysis 5: Comparison: Group 1: Immediate ART and Placebo Infusion vs Group 2: Immediate ART and VRC01 Infusion; Comparison of change in CD4+ T cells in Groups 1 and 2 from Baseline to Day 168; Test type: Superiority; p > .999, Wilcoxon (Mann-Whitney); Comparison of change in CD4+ T cells in Groups 1 and 2 from Baseline to Day 168 p-value calculated using 10,000 bootstrapped samples
Statistical Analysis 6: Comparison: Group 1: Immediate ART and Placebo Infusion vs Group 3: Immediate VRC01 Infusion and Subsequent ART; Comparison of change in CD4+ T cells in Groups 1 and 3 from Baseline to Day 168 p-value calculated using 10,000 bootstrapped samples; Test type: Superiority; p > .999, Wilcoxon (Mann-Whitney); Comparison of change in CD4+ T cells in Groups 1 and 3 from Baseline to Day 168 p-value calculated using 10,000 bootstrapped samples

12. Secondary Outcome: Measurement of VRC01 Levels in Peripheral Blood
Time Frame: Measured through Week 24
Population: The analysis population for this outcome is defined as those in the virologic population who have available samples for measuring the amount of VRC01 in the peripheral compartment. Some participants did not have samples available for the PK analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1: Immediate ART and Placebo Infusion | Group 2: Immediate ART and VRC01 Infusion | Group 3: Immediate VRC01 Infusion and Subsequent ART
Number analyzed (Participants) | 8 | 8 | 8
ng/mL
  Day 1 (Pre): number analyzed (Participants) | 8 | 8 | 7
  Day 1 (Pre) | 0 (0) | 0 (0) | 0 (0)
  Day 1 (Post): number analyzed (Participants) | 3 | 3 | 4
  Day 1 (Post) | 0 (0) | 1136.667 (303.078) | 741.250 (458.083)
  Day 3: number analyzed (Participants) | 8 | 8 | 7
  Day 3 | 0 (0) | 276.813 (81.678) | 259.600 (90.044)
  Day 7: number analyzed (Participants) | 8 | 8 | 7
  Day 7 | 0 (0) | 169.288 (46.161) | 156.043 (51.723)
  Day 14 | 0 (0) | 91.275 (27.295) | 87.750 (32.660)
  Day 21: number analyzed (Participants) | 6 | 6 | 6
  Day 21 | 0 (0) | 58.583 (17.117) | 47.717 (20.103)
  Day 28 | 0 (0) | 37.438 (19.377) | 32.850 (16.682)
  Day 56: number analyzed (Participants) | 8 | 8 | 6
  Day 56 | 0 (0) | 13.800 (16.716) | 7.933 (8.500)
  Day 168: number analyzed (Participants) | 8 | 7 | 6
  Day 168 | 0 (0) | 0 (0) | 3.350 (8.206)
Statistical Analysis 1: Comparison: Group 2: Immediate ART and VRC01 Infusion vs Group 3: Immediate VRC01 Infusion and Subsequent ART; Test type: Superiority; p = .8629, Wilcoxon (Mann-Whitney) — Multiple comparisons are not required

ADVERSE EVENTS:
Time Frame: Adverse event data are collected through 175 days after study agent administration.
Description: MedDRA version 21.2 was used. The site clinical research team will ascertain accurate recording of AEs on a daily basis. The clinical investigators will monitor and analyze study data as they become available and will make determinations regarding the severity of the adverse experiences and their relation to study product.
Arm/Group | Group 1: Immediate ART and Placebo Infusion | Group 2: Immediate ART and VRC01 Infusion | Group 3: Immediate VRC01 Infusion and Subsequent ART
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/8 | 1/8
Other Adverse Events (participants affected / at risk) | 8/8 | 7/8 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Immediate ART and Placebo Infusion (N=8) | Group 2: Immediate ART and VRC01 Infusion (N=8) | Group 3: Immediate VRC01 Infusion and Subsequent ART (N=8)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0
Anal fistula repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Immediate ART and Placebo Infusion (N=8) | Group 2: Immediate ART and VRC01 Infusion (N=8) | Group 3: Immediate VRC01 Infusion and Subsequent ART (N=8)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anorectal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (6) | 1 (3) | 2 (3)
Oral mucosa haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (3)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2)
Malaise (General disorders) | 2 (3) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Syphilis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urethritis gonococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (4) | 4 (6) | 4 (8)
Aspartate aminotransferase increased (Investigations) | 5 (6) | 4 (5) | 4 (6)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (6) | 3 (3) | 2 (3)
Headache (Nervous system disorders) | 3 (6) | 3 (4) | 5 (6)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Anal fistula repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Rhinoplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT02591420/Prot_SAP_000.pdf